CLINICAL TRIAL: NCT03048266
Title: Metabolomics and Genetic Diagnosing Pancreatic Neuroendocrine Tumors in Multiple Endocrine Neoplasia Type 1 Patients
Brief Title: Metabolomics and Genetic Diagnosing Pancreatic Neuroendocrine Tumors in MEN1 Patients
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA15-0822
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Multiple Endocrine Neoplasia
Keywords: Multiple endocrine neoplasia; MEN1; Aggressive pancreatic neuroendocrine tumors; PNET; Non-aggressive pancreatic neuroendocrine tumors; Metabolomics; Genetics; Biomarkers
MeSH Terms: conditions — Multiple Endocrine Neoplasia; Neuroectodermal Tumors, Primitive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MEN1 Patients Who Have Developed Aggressive PNETs-Cases
- MEN1 Patients Who Have Developed Non-Aggressive PNETs-Controls

SUMMARY:
Objectives:

The aim of the present study is to assess the significance of metabolomics and genetics in diagnosing and survival evaluation for pNET in the periodic follow-up of MEN1 patients.

Aim 1: To evaluate the relationship of serum global metabolic profiles with subsequent development of aggressive PNET and evaluate patients survival in a nested case-control study of MEN1 patients who have developed aggressive PNETs (cases) and MEN1 patients who have developed non-aggressive PNETs (controls).

Aim 2: Validate the top serum metabolites identified from Aim 1 in MEN1 patients who have developed aggressive PNETs and MEN1 patients who have developed non-aggressive PNETs, using a targeted metabolomics approach.

Aim 3: Prospectively identify the potential miRNA biomarkers of serum with miRNA sequencing in MEN1 patients who have developed aggressive PNETs (cases) and MEN1 patients who have developed non-aggressive PNETs (controls).

Aim 4: Validate the potential miRNA biomarkers identified from Aim 1 in MEN1 patients who have developed aggressive PNETs and in MEN1 patients who have developed non-aggressive PNETs, using a targeted qRT-PCR approach (in serums), as well as to see the relationship of potential miRNA biomarkers with patients survival.

ELIGIBILITY:
Inclusion Criteria:

1. The study will include all patients with a confirmed MEN1 diagnosis (clinical, genetic or familial criteria).
2. No prior history of PNET.

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study subjects identified from a cohort of MEN1 patients. These patients had previously consented to collection of clinical data, blood, and parathyroid tissue for research purposes at MD Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 629 (Estimated)
Dates: Start 2015-11-05 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Relationship of Serum Global Metabolic Profiles with Subsequent Development of Aggressive PNET | 10 years
  Review of samples from 50 cases (aggressive PNET) and 50 controls (non-aggressive PNET).

SECONDARY OUTCOMES:
Prediction of Occurrence of Aggressive PNET among MEN1 Patients by Examining Patterns of Serum Metabolic Biomarkers | 10 years
  Advanced metabolomics technology used to demonstrate that various patterns of serum metabolic biomarkers can predict the occurrence of aggressive PNET among MEN1 patients.
Prospectively Identify Potential miRNA Biomarkers of Serum with miRNA Sequencing in MEN1 Patients Who Have Developed Aggressive PNETs (Cases) and MEN1 Patients Who Have Developed Non-Aggressive PNETs (Controls) | 10 years
  The levels of miRNA in each group defined as mean ±SD. One-way ANOVA used to identify possible associations between miRNA concentrations and clinicopathological features of aggressive patients.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy D. Perrier, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org